CLINICAL TRIAL: NCT05985317
Title: Evaluation of Collagen Versus Platelet Rich Fibrin Membrane on the Osteogenic Potential of Bone Marrow Aspirate Concentrate (BMAC) for Lateral Sinus Floor Augmentation : A Randomized Clinical Trial.
Brief Title: Effect of Collagen Versus PRF on BMA Osteogenic Potential
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Walaa Kadry, Lecturer of oral and Maxillofacial Surgery, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: The membrane effect on the BM
Record Dates: First submitted 2023-07-23; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Bone Loss, Alveolar
MeSH Terms: conditions — Alveolar Bone Loss

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Collagen membrane covering BMAC loaded on bovine graft (Active Comparator): Collagen membrane will be used to BMAC loaded on bovine graft . Variables include assessment of the osteogenic potential In terms of bone density measurements of graft immediate and 4 months Postoperative
  Interventions: Procedure: Collagen membrane over BMAC/bovine graft in sinus lift
- PRF membrane covering BMAC loaded on bovine graft (Active Comparator): Platelet rich fibrin membrane will be used to BMAC loaded on bovine graft . Variables include assessment of the osteogenic potential In terms of bone density measurements of graft immediate and 4 months Postoperative
  Interventions: Procedure: PRF membrane over BMAC/bovine graft in sinus lift

INTERVENTIONS:
Procedure: Collagen membrane over BMAC/bovine graft in sinus lift — Collagen membrane to cover BMAC/bovine graft in sinus lift and evaluation of its effect on osteogenic potential of BMAC in sinus lift procedure
  Arms: Collagen membrane covering BMAC loaded on bovine graft
Procedure: PRF membrane over BMAC/bovine graft in sinus lift — PRF membrane to cover BMAC/bovine graft in sinus lift and evaluation of its effect on osteogenic potential of BMAC in sinus lift procedure
  Arms: PRF membrane covering BMAC loaded on bovine graft

SUMMARY:
Utilization of collagen vs PRF membrane over the graft following sinus lift procedure and before suturing

DETAILED DESCRIPTION:
Assessment of the effect of membrane overlying bone marrow aspirate concentrate - bovine graft mixture in sinus lift procedure

ELIGIBILITY:
Inclusion Criteria:

* Patients who has as deficient as 4 mm vertical bone height in posterior maxilla that need bone augmentation before delayed implant placement.
* Highly motivated patients
* Age more than 18 years

Exclusion Criteria:

* Patients suffering from any systemic disease or those under any medication that may interfere with normal bone healing.
* Patients suffering from any sinus pathosis.
* Patients with conditions that could potentially compromise Bone Marrow ( BM)quality, including history of hematologic malignancy, current chemotherapy, BM suppressive and anti-platelet medications, previous BM Aspiration, or acute illness.
* Heavy smoker (> 20 cigarettes daily)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2 (Estimated)
Dates: Start 2023-01-25 (Actual); Primary Completion 2023-08-30 (Estimated); Study Completion 2023-08-30 (Estimated)

PRIMARY OUTCOMES:
Radiographic Bone density assessment | 4 months ( immediate - 4 months postoperative)
  Bone density measurements on Cone beam CT/CBCT immediate and 4 months radiographic density measurements in haunsfield units, immediate and 4 months postoperative

SECONDARY OUTCOMES:
Radiographic Bone height assessment | 4 months ( immediate - 4 months postoperative)
  Assessment of bone hight on CBCT, mmediate and at 4 months postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Eman Said, Study Director — Lecturer at Faculty of Dentistry, Cairo University
Locations (1):
- Faculty of Dentistry, Cairo University, Cairo, Egypt